CLINICAL TRIAL: NCT02093273
Title: Phase II, Randomized, Double Blind, Prospective Intervention Study to Evaluate the Immunogenicity and Safety Profile of tOPV (Bio Farma) With Different Batch Numbers in Indonesian Infants
Brief Title: Evaluation on Immunogenicity and Safety Profile of Trivalent OPV (tOPV Bio Farma)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OPV 0213
Record Dates: First submitted 2014-03-19; First posted 2014-03-20 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: tOPV; Antibody response; Safety
MeSH Terms: interventions — Poliovirus Vaccine, Oral

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tOPV commercial batch (Bio Farma) (Active Comparator): tOPV (Bio Farma) one dose correspond to 2 drops (0.1ml)
  Interventions: Biological: tOPV commercial batch
- tOPV pilot batch (Experimental): tOPV (Bio Farma), one dose correspond to 2 drops (0.1ml)
  Interventions: Biological: tOPV pilot batch

INTERVENTIONS:
Biological: tOPV pilot batch — the tOPV vaccine is given orally
  Other Names: tOPV (Bio Farma)
  Arms: tOPV pilot batch
Biological: tOPV commercial batch — tOPV vaccine is given orally
  Other Names: tOPV (Bio Farma)
  Arms: tOPV commercial batch (Bio Farma)

SUMMARY:
The objective of this study is to compare the antibody response 30 days after two doses of t OPV

DETAILED DESCRIPTION:
The trial design is phase II, randomized, double blind, prospective intervention study. The subject study are 240 healthy, full term, newborn infants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, full term, newborns infants
* newborn residing within a relatively short and easily accessible distance A(<30km) from the study clinic(s) and not planning to travel away during the entire study period
* Infant born after 37 weeks of pregnancy
* Infant weighing 2.5kg or more at birth (birth weight >= 2.5kg)
* Healthy newborns, with no history of asphyxia or meconium aspiration
* Father, mother or legally acceptable representative properly informed about the study and having signed the informed consent form.
* Parents will commit themselves to comply with the indications of the investigator and with the schedule of the trial
* Mother at least elementary school graduate

Exclusion Criteria:

* Child concomitantly enrolled or scheduled to be enrolled in another trial
* Known history of congenital or acquired immunodeficiency (including HIV infection)
* Evolving moderate or severe illness, especially infectious diseases or fever (axillary temperature >=37.5oC
* Newborns requiring hospitalization at birth
* Infant immunized with non-scheduled OPV or IPV during trial

Ages: 1 Minute to 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2013-05; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To compare the antibody response 30 days after two doses of tOPV | 30 days
  antibody titer to Polio

SECONDARY OUTCOMES:
To asses and compare the safety of tOPV | 30 days
  Data collection of local and systemic reaction after immunization

OTHER OUTCOMES:
To describe the antibody response after two doses of tOPV | 30 days
  Measurement of titer antibody

CONTACTS AND LOCATIONS:
Overall Officials: Eddy Fadlyana, MD, Principal Investigator — Department of Child Health of Medicine Padjadjaran University
Locations (4):
- Indonesia (4):
  - Garuda Primary Health Center, Bandung, West Java
  - Ibrahim Adjie Primary Health Centre, Bandung, West Java
  - Padasuka Primary Health Centre, Bandung, West Java
  - Puter Primary Health Centre, Bandung, West Java